CLINICAL TRIAL: NCT04575545
Title: Prevalence of COVID-19 Infection in a Cohort of Patient Infected by the HIV and Patients Taking PrEP Pre-exposure Prophylaxis
Brief Title: Prevalence of COVID-19 Infection in a Cohort of Patients Infected by the HIV and Patients Taking PrEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02018-31
Record Dates: First submitted 2020-10-02; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Virus-HIV
MeSH Terms: conditions — COVID-19; Acquired Immunodeficiency Syndrome | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV positive patients
  Interventions: Diagnostic Test: Serology test for COVID-19
- Patients taking PrEP
  Interventions: Diagnostic Test: Serology test for COVID-19

INTERVENTIONS:
Diagnostic Test: Serology test for COVID-19 — ELISA test

SUMMARY:
The purpose of the study is to assess seroprevalence of COVID-19 infection in a cohort of HIV + patients and in a cohort of patients taking PrEP by emtricitabine / tenofovir.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* patients infected by the HIV on treatment
* patients taking PreP (Pre-exposure prophylaxis (PrEP))
* Being affiliated with or benefiting from a social security scheme

Exclusion Criteria:

* Subject to a measure for the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients infected by the HIV on treatment and patients taking PreP
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
% of patients with positive serological tests for covid-19 | 3 months

SECONDARY OUTCOMES:
Presence and quantification of CD4 / CD8 reactivity to COVID-19 epitopes in patient with positive and negative serological tests for covid-19 | 3 months
  % of anti-covid positive cells

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PHILIBERT, Principal Investigator — Hôpital Europeen Marseille
Locations (1):
- BENNANI, Marseille, France